CLINICAL TRIAL: NCT01864304
Title: Characterization of Fat Distribution and Glucose Metabolism in Individuals With and Without Williams Syndrome
Brief Title: Fat Distribution and Glucose Metabolism in Williams Syndrome
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Takara Stanley, M.D., Assistant Pediatrician, Massachusetts General Hospital
Other Study IDs: 2013P000068
Record Dates: First submitted 2013-05-10; First posted 2013-05-29 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Williams Syndrome
Keywords: Williams Syndrome
MeSH Terms: conditions — Williams Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Williams Syndrome: Children and adults with Williams Syndrome
- Control Group: Controls will be recruited in 2 ways: 1) a gender matched and age- and BMI-similar control for each WS patient, and, 2) sibling controls when available

SUMMARY:
Williams Syndrome (WS) is a genetic syndrome with features that may include vascular stenoses, neuro-developmental changes, and a variety of endocrine and metabolic abnormalities, including impaired glucose metabolism and abnormal body composition. Approximately 75% of adults with WS have impaired glucose tolerance or diabetes on oral glucose tolerance testing (OGTT). In addition, clinical observations and preliminary data suggest increased overall body fat in these individuals, as well as a relative increase in fat deposition in the lower extremities. However, glucose and lipid metabolism in WS remain incompletely characterized. The purpose of the current study is to carefully describe glucose metabolism and lipid parameters in people with WS.

ELIGIBILITY:
Inclusion Criteria

1. M or F age 14-70yo
2. Diagnosis of WS confirmed by FISH or chromosomal microarray (WS only)
3. Availability of a parent or guardian to participate in the consent process (all WS, and controls <18yo)

Exclusion Criteria

1. History of weight loss surgery or liposuction
2. Use of weight-lowering drugs
3. Positive urine pregnancy test (females only)
4. Obesity or abnormal fat distribution due to a known secondary cause (except WS) such as Cushing syndrome, HIV-infection, etc.
5. Known diabetes will preclude administration of the OGTT but not participation in other aspects of the study.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with Williams Syndrome (WS), and "control" individuals without WS.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
2-hour glucose | Baseline
  Blood glucose concentration two hours after drinking a sugary drink (oral glucose tolerance test)

SECONDARY OUTCOMES:
Percent body fat | Baseline
  percent body fat as measured by whole body dual-energy xray absorptiometry (DXA) scanning
Low-density lipoprotein cholesterol (LDL) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Takara Stanley, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States